CLINICAL TRIAL: NCT00878644
Title: Therapeutic Hypothermia After Pediatric Cardiac Arrest (Out of Hospital)
Brief Title: Therapeutic Hypothermia to Improve Survival After Cardiac Arrest in Pediatric Patients-THAPCA-OH [Out of Hospital] Trial
Acronym: THAPCA-OH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frank W. Moler, M.D, M.S, Professor of Pediatrics, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 619; U01HL094339 (NIH)
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-07

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest; Cardiopulmonary Arrest; Pediatric Cardiac Arrest; VABS; Vineland Adaptive Behavior Survey; POPC/PCPC; hypoxic-ichemic encephalopathy
MeSH Terms: conditions — Heart Arrest | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic Hypothermia (Experimental): Participants will receive therapeutic hypothermia after experiencing cardiac arrest.
  Interventions: Procedure: Therapeutic Hypothermia
- Therapeutic Normothermia (Active Comparator): Participants will receive therapeutic normothermia after experiencing cardiac arrest.
  Interventions: Other: Therapeutic Normothermia

INTERVENTIONS:
Procedure: Therapeutic Hypothermia — Participants who are assigned to receive hypothermia will be cooled to a target temperature of 33º C plus or minus 1º C (32 to 34º C). This temperature will be maintained for 48 hours (2 days) and then participants will be warmed to a target temperature of 36.75º C plus or minus 0.75º C (36 to 37.5º C). This temperature will be maintained until 120 hours (5 days) after the cardiac arrest.
  Arms: Therapeutic Hypothermia
Other: Therapeutic Normothermia — Participants who are assigned to receive therapeutic normothermia will have their temperature maintained at 36.75º C plus or minus 0.75º C (36° to 37.5º C) for 120 hours (5 days) after the cardiac arrest.
  Arms: Therapeutic Normothermia

SUMMARY:
Cardiac arrest is a sudden, unexpected loss of heart function. Therapeutic hypothermia, in which the body's temperature is lowered and maintained several degrees below normal for a period of time, has been used to successfully treat adults who have experienced cardiac arrest. This study will evaluate the efficacy of therapeutic hypothermia at increasing survival rates and reducing the risk of brain injury in infants and children who experience a cardiac arrest while out of the hospital.

DETAILED DESCRIPTION:
Cardiac arrest occurs when the heart suddenly stops beating and blood flow to the body is halted. It can occur while people are in the hospital because of a medical condition, or while people are out of the hospital as a result of an accident or other causes. Cardiac arrest is a serious event that is associated with high rates of death and long-term disability. When a person experiences cardiac arrest, insufficient amount of blood flow and oxygen can result in brain injury.

Therapeutic hypothermia is a therapy that involves a controlled lowering of the body temperature and then maintenance of this lower temperature for a period of time. The treatment may result in reduced brain injury. Therapeutic hypothermia has been successfully used in adults who experience cardiac arrest to improve survival rates and health outcomes, and it has also been studied in newborn infants who have suffered from perinatal asphyxia. The purpose of this study is to evaluate the efficacy of therapeutic hypothermia at improving survival rates and reducing brain injury in infants and children who experience cardiac arrest while out of the hospital.

Study researchers will conduct this study in collaboration with the following two pediatric clinical research networks: the Pediatric Emergency Care Applied Research Network (PECARN), funded by the Emergency Medical Services for Children (EMSC) program, and the National Institute of Child Health and Human Development (NICHD) Collaborative Pediatric Critical Care Research Network (CPCCRN).

The study will enroll infants and children who have suffered a cardiac arrest while out of the hospital. Randomization must occur within 6 hours of return of spontaneous circulation. Participants will be randomly assigned to receive either therapeutic hypothermia or therapeutic normothermia. Participants receiving therapeutic hypothermia will have their body temperature reduced to between 32 to 34° Celsius (C) and will remain at this temperature for 2 days. Their body temperature will then be slowly increased to the normal temperature of 36 to 37.5° C, which will be maintained until 5 days after the cardiac arrest. Participants receiving therapeutic normothermia will have their normal temperature maintained between 36 to 37.5° C for 5 days after the cardiac arrest. Special temperature control blankets will be placed to maintain body temperature in the assigned range. After 5 days, each participant's temperature will be managed by their medical care team.

While participants are in the hospital, they will undergo frequent blood and urine collections, chest x-rays, and temperature measurements; parents of participants will complete questionnaires. When participants are ready to leave the hospital, study researchers will perform a physical and functional assessment. Twenty-eight days after the cardiac arrest, researchers will contact parents of participants to gather information on the participants' health and medical condition. At Months 3 and 12, a child development expert will contact parents to gather medical information. At Month 12, participants will attend a study visit for a neurologic examination and testing with a psychologist trained in rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffered cardiac arrest requiring chest compressions for at least 2 minutes (120 seconds) with ROSC/ROC; AND
* Age greater than 48 hours (with a corrected gestational age of at least 38 weeks) and less than 18 years; AND
* Patient requires continuous mechanical ventilation; AND
* The cardiac arrest was unplanned (i.e., not part of cardiac surgical procedure)

Exclusion Criteria:

* The parent or legal guardian does not speak English or Spanish (the only two languages in which VABS II is standardized)
* Randomization is impossible within six hours of ROSC; OR
* Patient is on extracorporeal membrane oxygenation (ECMO) when arrest occurs; OR
* Continuous infusion of epinephrine or norepinephrine at very high doses (≥2 ug/kg/minute) received immediately prior to randomization; OR Glasgow Coma Scale motor response of five (localizing pain or for infants less than two years, withdraws to touch) or six (obeys commands, or for infants, normal spontaneous movement) prior to randomization; OR
* History of a prior cardiac arrest with chest compressions for at least two minutes during the current hospitalization but outside the 6 hour window for randomization; OR
* Pre-existing terminal illness with life expectancy < 12 months; OR
* Lack of commitment to aggressive intensive care therapies including do not resuscitate orders and other limitations to care; OR
* Cardiac arrest was associated with severe brain, thoracic, or abdominal trauma; OR
* Active and refractory severe bleeding prior to randomization; OR
* Near drowning in ice water with patient core temperature ≤32 °C on presentation; OR
* Patient is pregnant; OR
* Patient participation in a concurrent interventional trial whose protocol, in the judgment of the THAPCA investigators, prevents effective application of one or both THAPCA therapeutic treatment arms, or otherwise significantly interferes with carrying out the THAPCA protocol; OR
* Patient is newborn with acute birth asphyxia; OR

  _ Patient cared for in a neonatal intensive care unit (NICU) after arrest (ie, would not be admitted to PICU); OR
* Patient has sickle cell anemia; OR
* Patient known to have pre-existing cryoglobulinemia; OR
* Central nervous system tumor with ongoing chemotherapy or radiation therapy; OR
* Chronic hypothermia secondary to hypovolemic, pituitary, or related condition for which body temperature is consistently below 37 °C ; OR progressive degenerative encephalopathy; OR
* Any condition in which direct skin surface cooling would be contraindicated, such as large burns, decubitus ulcers, cellulitis, or other conditions with disrupted skin integrity (NOTE: patients with open chest CPR should be included but placement of cooling mattresses will be modified as needed); OR
* Previous enrollment in the THAPCA Trials.

Ages: 48 Hours to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 295 (Actual)
Dates: Start 2009-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank W Moler, MD, MS, Principal Investigator — University of Michigan; Michael Dean, MD, MBA, Principal Investigator — University of Utah
Locations (34):
- United States (33):
  - The Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of Arizona at Tucson, Tucson, Arizona
  - Loma Linda University Children's Hospital, Loma Linda, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California San Francisco, San Francisco, California
  - Children's Hospital of Denver/University of Colorado, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Atlanta/Emory University, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Kosair Children's Hospital, Louisville, Kentucky
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - University of Michigan, Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Children's Hospital of New York - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke Children's Hospital, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Rainbow Babies and Children, Cleveland, Ohio
  - Nationwide Children's Hospital in Columbus, Columbus, Ohio
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philidelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - LeBonheur Children's Hospital - University of Tennessee at Memphis, Memphis, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - University of Texas Health Sciences Center of San Antonio, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Seatlle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin/Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meert KL, Donaldson A, Nadkarni V, Tieves KS, Schleien CL, Brilli RJ, Clark RS, Shaffner DH, Levy F, Statler K, Dalton HJ, van der Jagt EW, Hackbarth R, Pretzlaff R, Hernan L, Dean JM, Moler FW; Pediatric Emergency Care Applied Research Network. Multicenter cohort study of in-hospital pediatric cardiac arrest. Pediatr Crit Care Med. 2009 Sep;10(5):544-53. doi: 10.1097/PCC.0b013e3181a7045c. PMID 19451846
- [Result] Moler FW, Meert K, Donaldson AE, Nadkarni V, Brilli RJ, Dalton HJ, Clark RS, Shaffner DH, Schleien CL, Statler K, Tieves KS, Hackbarth R, Pretzlaff R, van der Jagt EW, Levy F, Hernan L, Silverstein FS, Dean JM; Pediatric Emergency Care Applied Research Network. In-hospital versus out-of-hospital pediatric cardiac arrest: a multicenter cohort study. Crit Care Med. 2009 Jul;37(7):2259-67. doi: 10.1097/CCM.0b013e3181a00a6a. PMID 19455024
- [Result] Moler FW, Donaldson AE, Meert K, Brilli RJ, Nadkarni V, Shaffner DH, Schleien CL, Clark RS, Dalton HJ, Statler K, Tieves KS, Hackbarth R, Pretzlaff R, van der Jagt EW, Pineda J, Hernan L, Dean JM; Pediatric Emergency Care Applied Research Network. Multicenter cohort study of out-of-hospital pediatric cardiac arrest. Crit Care Med. 2011 Jan;39(1):141-9. doi: 10.1097/CCM.0b013e3181fa3c17. PMID 20935561
- [Result] Moler FW, Silverstein FS, Holubkov R, Slomine BS, Christensen JR, Nadkarni VM, Meert KL, Clark AE, Browning B, Pemberton VL, Page K, Shankaran S, Hutchison JS, Newth CJ, Bennett KS, Berger JT, Topjian A, Pineda JA, Koch JD, Schleien CL, Dalton HJ, Ofori-Amanfo G, Goodman DM, Fink EL, McQuillen P, Zimmerman JJ, Thomas NJ, van der Jagt EW, Porter MB, Meyer MT, Harrison R, Pham N, Schwarz AJ, Nowak JE, Alten J, Wheeler DS, Bhalala US, Lidsky K, Lloyd E, Mathur M, Shah S, Wu T, Theodorou AA, Sanders RC Jr, Dean JM; THAPCA Trial Investigators. Therapeutic hypothermia after out-of-hospital cardiac arrest in children. N Engl J Med. 2015 May 14;372(20):1898-908. doi: 10.1056/NEJMoa1411480. Epub 2015 Apr 25. PMID 25913022
- [Derived] Harhay MO, Blette BS, Granholm A, Moler FW, Zampieri FG, Goligher EC, Gardner MM, Topjian AA, Yehya N. A Bayesian Interpretation of a Pediatric Cardiac Arrest Trial (THAPCA-OH). NEJM Evid. 2023 Jan;2(1):EVIDoa2200196. doi: 10.1056/EVIDoa2200196. Epub 2022 Dec 14. PMID 38320098
- [Derived] Siddique J. Bayesian (re)-Analyses of Clinical Trial Data. NEJM Evid. 2023 Jan;2(1):EVIDe2200297. doi: 10.1056/EVIDe2200297. Epub 2022 Dec 27. PMID 38320013
- [Derived] Slomine BS, Silverstein FS, Page K, Holubkov R, Christensen JR, Dean JM, Moler FW; Therapeutic Hypothermia after Pediatric Cardiac Arrest (THAPCA) Trial Investigators. Relationships between three and twelve month outcomes in children enrolled in the therapeutic hypothermia after pediatric cardiac arrest trials. Resuscitation. 2019 Jun;139:329-336. doi: 10.1016/j.resuscitation.2019.03.020. Epub 2019 Mar 26. PMID 30922934
- [Derived] Moler FW, Silverstein FS, Nadkarni VM, Meert KL, Shah SH, Slomine B, Christensen J, Holubkov R, Page K, Dean JM; THAPCA Trial Investigators. Pediatric out-of-hospital cardiac arrest: Time to goal target temperature and outcomes. Resuscitation. 2019 Feb;135:88-97. doi: 10.1016/j.resuscitation.2018.12.012. Epub 2018 Dec 17. PMID 30572071
- [Derived] Ichord R, Silverstein FS, Slomine BS, Telford R, Christensen J, Holubkov R, Dean JM, Moler FW; THAPCA Trial Group. Neurologic outcomes in pediatric cardiac arrest survivors enrolled in the THAPCA trials. Neurology. 2018 Jul 10;91(2):e123-e131. doi: 10.1212/WNL.0000000000005773. Epub 2018 Jun 8. PMID 29884735
- [Derived] Meert K, Telford R, Holubkov R, Slomine BS, Christensen JR, Dean JM, Moler FW; Therapeutic Hypothermia after Paediatric Cardiac Arrest (THAPCA) Trial Investigators. Exploring the safety and efficacy of targeted temperature management amongst infants with out-of-hospital cardiac arrest due to apparent life threatening events. Resuscitation. 2016 Dec;109:40-48. doi: 10.1016/j.resuscitation.2016.09.026. Epub 2016 Oct 11. PMID 27737774
- [Derived] Slomine BS, Silverstein FS, Christensen JR, Holubkov R, Page K, Dean JM, Moler FW; THAPCA Trial Group. Neurobehavioral Outcomes in Children After Out-of-Hospital Cardiac Arrest. Pediatrics. 2016 Apr;137(4):e20153412. doi: 10.1542/peds.2015-3412. Epub 2016 Mar 3. PMID 26940987
- [Derived] Holubkov R, Clark AE, Moler FW, Slomine BS, Christensen JR, Silverstein FS, Meert KL, Pollack MM, Dean JM. Efficacy outcome selection in the therapeutic hypothermia after pediatric cardiac arrest trials. Pediatr Crit Care Med. 2015 Jan;16(1):1-10. doi: 10.1097/PCC.0000000000000272. PMID 25268768
- [Derived] Moler FW, Silverstein FS, Meert KL, Clark AE, Holubkov R, Browning B, Slomine BS, Christensen JR, Dean JM. Rationale, timeline, study design, and protocol overview of the therapeutic hypothermia after pediatric cardiac arrest trials. Pediatr Crit Care Med. 2013 Sep;14(7):e304-15. doi: 10.1097/PCC.0b013e31828a863a. PMID 23842585
- [Derived] Pemberton VL, Browning B, Webster A, Dean JM, Moler FW. Therapeutic hypothermia after pediatric cardiac arrest trials: the vanguard phase experience and implications for other trials. Pediatr Crit Care Med. 2013 Jan;14(1):19-26. doi: 10.1097/PCC.0b013e31825b860b. PMID 23295834

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia
Started | 155 | 140
Completed | 151 | 136
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia | Total
Number analyzed (Participants) | 155 | 140 | 295
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 2.1 [0.6 to 10.1] | 1.6 [0.4 to 7.0] | 2.0 [0.5 to 8.7]
Age, Customized [Count of Participants; unit: Participants]
  Age Category: < 2 yr | 76 | 73 | 149
  Age Category: 2 - <12 yr | 48 | 45 | 93
  Age Category: 12 - 17 yr | 31 | 22 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 46 | 99
  Male | 102 | 94 | 196

OUTCOME MEASURES:

1. Primary Outcome: Survival With Good Neurobehavioral Outcome
Description: Survival at one-year anniversary of cardiac arrest, with a standardized VABS-II score of 70 or greater per evaluation performed at any time from 30 days prior to until 183 days after the one-year anniversary of cardiac arrest.
Time Frame: Survival was assessed at one-year anniversary of cardiac arrest; among survivors at this one-year anniversary, the VABS-II valid assessment window ranged from 30 days prior to until 183 days after the one-year anniversary date.
Population: Subjects with baseline VABS-II >= 70, OR unavailable baseline VABS-II but Pediatric Overall Performance Category (POPC) score and Pediatric Cerebral Overall Performance Category (PCPC) both reflecting none or mild disability (1 or 2), are eligible for the primary analysis. Population is analysis-eligible patients with available primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia
Number analyzed (Participants) | 138 | 122
Participants
  Alive with VABS-II >=70 at 1 year | 27 | 15
  Died or Alive with VABS-II <70 at 1 year | 111 | 107
Statistical Analysis 1: Comparison: Therapeutic Hypothermia vs Therapeutic Normothermia; Test type: Superiority; p = 0.14, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test was used adjusting for age category at time of randomization (<2 years, 2 to <12 years, or >=12 years); Risk Difference (RD) = 7.3, 95% CI 2-sided [-1.5 to 16.1]

2. Secondary Outcome: Survival
Description: Survival at one year after cardiac arrest
Time Frame: Measured at one-year anniversary of cardiac arrest.
Population: All randomized patients with available vital status (alive or deceased) at one year after cardiac arrest.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia
Number analyzed (Participants) | 151 | 136
Participants
  Alive at 1 year | 57 | 39
  Died at 1 year | 94 | 97
Statistical Analysis 1: Comparison: Therapeutic Hypothermia vs Therapeutic Normothermia; Test type: Superiority; p = 0.13, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 9.1, 95% CI 2-sided [-1.8 to 19.9]

3. Secondary Outcome: Change in Neurobehavioral Function From Pre-cardiac Arrest to 12 Months Post-cardiac Arrest
Description: Change in VABS-II score from baseline to one year, with death at 1 year treated as worst possible outcome, and lowest possible VABS-II score at one year (regardless of baseline VABS-II score) treated as the second worst possible outcome.
Time Frame: as for outcome 1
Population: All randomized subjects with available data for this outcome (this implies a child must be either dead at 1 year, have the lowest possible value for the VABS-II score at 1 year, or if neither of these two criteria applies, must have both baseline VABS-II and 1-year VABS-II scores available to allow calculation of change in VABS-II score)
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia
Number analyzed (Participants) | 151 | 134
Participants
  Dead at 1 year | 94 | 97
  Lowest possible VABS-II at 1 year | 6 | 1
  1-year decrease in VABS-II >30 points | 19 | 15
  1-year decrease in VABS-II 16-30 points | 11 | 4
  1-year decrease in VABS-II <=15 points or improved | 21 | 17
Statistical Analysis 1: Comparison: Therapeutic Hypothermia vs Therapeutic Normothermia; Test type: Superiority; p = 0.13, Stratified Mann-Whitney Test; Test stratified by age category (<2 years, 2 to <12 years, or >=12 years), for continuous (NOT categorized as reported above) 1-year change in VABS-II; As the (nonparametric) comparison treated 1-year deaths as worst possible outcomes and worst possible 1-year VABS-II as next worst possible outcomes, using change in VABS-II for other participants alive at 1 year, no relevant estimation of effect size is possible for this secondary outcome

4. Secondary Outcome: Neuropsychological Scores (for Participants That Survive)
Description: Functioning, as assessed by the Mullen Early Learning Composite (for children age < 5 years 9 months) or by the 2-subset version of the Wechsler Abbreviated Scale of Intelligence (WASI). As these two function measures are scaled in the same fashion, the two age groups are combined.
Time Frame: Measured at Month 12
Population: Randomized children alive at one year with neuropsychological score available.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia
Number analyzed (Participants) | 52 | 35
Participants
  Lowest possible score | 27 | 17
  <70 (well below average) | 7 | 8
  70 - 84 (below average) | 5 | 6
  85 - 115 (average) | 8 | 2
  >115 (above average) | 5 | 2
Statistical Analysis 1: Comparison: Therapeutic Hypothermia vs Therapeutic Normothermia; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney); Test used the continuous (NOT categorized as reported above) neuropsychological scores, with "Lowest Possible Score" treated as lowest possible value

ADVERSE EVENTS:
Time Frame: For all-cause mortality, results reflect vital status at 12 months. Serious adverse events and other (not serious) adverse events were collected for 14 days after treatment was initiated.
Description: For adverse events, denominators reflect Safety Population of those patients receiving each treatment. Therefore, denominators are 153 patients receiving Therapeutic Hypothermia and 139 patients receiving Therapeutic Normothermia. For all-cause mortality, denominators additionally include only those with known 12-month vital status.
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia
All-Cause Mortality (participants affected / at risk) | 92/149 | 96/135
Serious Adverse Events (participants affected / at risk) | 98/153 | 102/139
Other Adverse Events (participants affected / at risk) | 145/153 | 124/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Hypothermia (N=153) | Therapeutic Normothermia (N=139)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bigeminy (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 3 (3) | 3 (3)
Cardiac arrest (Cardiac disorders) | 5 (6) | 9 (10)
Cardiac failure (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac failure aggravated (Cardiac disorders) | 0 (0) | 2 (2)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Torsades de pointes (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 2 (2)
Anisocoria (Eye disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multi organ failure (General disorders) | 0 (0) | 1 (1)
Multi-organ disorder (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 1 (1)
Multiorgan failure (General disorders) | 1 (1) | 0 (0)
Multiple organ failure (General disorders) | 2 (2) | 2 (2)
Shivering (General disorders) | 1 (1) | 0 (0)
Sudden infant death syndrome (General disorders) | 1 (1) | 0 (0)
Liver failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Candida albicans infection (Infections and infestations) | 0 (0) | 1 (1)
Infection pseudomonas aeruginosa (Infections and infestations) | 0 (0) | 1 (2)
Respiratory infection (Infections and infestations) | 4 (4) | 5 (6)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary infection (Infections and infestations) | 2 (2) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Brain stem herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac output decreased (Investigations) | 1 (1) | 0 (0)
HIE (Investigations) | 2 (2) | 1 (1)
QT interval prolonged (Investigations) | 1 (1) | 0 (0)
Sputum culture positive (Investigations) | 0 (0) | 1 (1)
Urine culture positive (Investigations) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Anoxic brain damage (Nervous system disorders) | 14 (14) | 14 (14)
Anoxic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Basal ganglia infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral edema (Nervous system disorders) | 13 (13) | 15 (15)
Cerebral infarct (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischemia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic brain damage (Nervous system disorders) | 10 (10) | 4 (4)
Hypoxic encephalopathy (Nervous system disorders) | 18 (18) | 21 (21)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Ischemia cerebral (Nervous system disorders) | 0 (0) | 2 (2)
Loss of gag reflex (Nervous system disorders) | 0 (0) | 1 (1)
Neurological status deterioration (Nervous system disorders) | 1 (1) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alkalosis respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pulmonary edema aggravated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory failure aggravated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cardiovascular collapse (Vascular disorders) | 1 (1) | 0 (0)
Circulatory failure (Vascular disorders) | 1 (1) | 0 (0)
DVT (Vascular disorders) | 1 (1) | 1 (1)
Hemodynamic instability (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 4 (4)
Ischemia (Vascular disorders) | 2 (2) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Hypothermia (N=153) | Therapeutic Normothermia (N=139)
Anemia (Blood and lymphatic system disorders) | 30 (32) | 18 (19)
Clotting (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulation disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 16 (16) | 9 (9)
DIC (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 9 (9) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Methemoglobinemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (16) | 2 (2)
2nd degree heart block (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Atrial arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bigeminy (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 12 (12) | 5 (5)
Bundle branch block (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 2 (2) | 1 (1)
Fibrosis myocardial (Cardiac disorders) | 0 (0) | 1 (1)
Junctional arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Junctional rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Mitral regurgitation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial depression (Cardiac disorders) | 2 (2) | 1 (1)
PVC's (Cardiac disorders) | 3 (3) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pneumopericardium (Cardiac disorders) | 2 (2) | 0 (0)
Premature ventricular contractions (Cardiac disorders) | 1 (1) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
SVT (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Stenosis pulmonic valve (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 7 (8)
Ventricular bigeminy (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 3 (3)
Hydrocele male (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear discharge (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2)
Diabetes insipidus (Endocrine disorders) | 16 (16) | 20 (20)
Anisocoria (Eye disorders) | 1 (1) | 1 (1)
Dilatation pupillary (Eye disorders) | 0 (0) | 1 (1)
Dilated pupils (Eye disorders) | 0 (0) | 1 (1)
Eye movement disorder (Eye disorders) | 1 (1) | 0 (0)
Fixed dilated pupils (Eye disorders) | 0 (0) | 1 (1)
Gaze palsy (Eye disorders) | 0 (0) | 1 (1)
Pupil fixed (Eye disorders) | 1 (1) | 0 (0)
Pupillary reaction slow (Eye disorders) | 0 (0) | 1 (1)
Retinal hemorrhage (Eye disorders) | 1 (1) | 3 (3)
Retinopathy hemorrhagic (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (2)
Bleeding mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloody stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel ischemia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Distended abdomen (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Emesis (Gastrointestinal disorders) | 4 (4) | 3 (3)
Esophageal tear (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fecal impaction (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI bleed (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gas (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal mucosal sloughing (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gum erosion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal edema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral discharge (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 9 (9) | 7 (7)
Pancreatitis aggravated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Saliva secretion excessive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stools watery (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swallowing difficult (Gastrointestinal disorders) | 1 (1) | 0 (0)
Swallowing disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
UGI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomited (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2)
Anasarca (General disorders) | 1 (1) | 3 (3)
Catheter related complication (General disorders) | 1 (1) | 0 (0)
Catheter site bleeding (General disorders) | 0 (0) | 2 (2)
Drug withdrawal syndrome (General disorders) | 3 (3) | 0 (0)
Edema (General disorders) | 7 (7) | 4 (4)
Edema abdomen (General disorders) | 1 (1) | 0 (0)
Edema extremity upper (General disorders) | 1 (1) | 0 (0)
Edema hands (General disorders) | 1 (1) | 0 (0)
Edema of extremities (General disorders) | 0 (0) | 1 (1)
Edema of lower extremities (General disorders) | 1 (1) | 2 (2)
Edema thigh (General disorders) | 1 (1) | 0 (0)
Edema trunk (General disorders) | 1 (1) | 0 (0)
Extravasation (General disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 16 (18) | 10 (10)
Generalized edema (General disorders) | 2 (2) | 1 (1)
Hand swelling (General disorders) | 1 (1) | 0 (0)
High temperature (General disorders) | 1 (1) | 0 (0)
Hyperpyrexia (General disorders) | 1 (2) | 0 (0)
Hyperthermia (General disorders) | 2 (2) | 2 (3)
Hypothermia (General disorders) | 1 (1) | 4 (4)
Infiltration intravenous injection (General disorders) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 2 (2) | 0 (0)
Infusion site infiltration (General disorders) | 1 (1) | 0 (0)
Intermittent fever (General disorders) | 1 (1) | 0 (0)
Leg edema (General disorders) | 1 (1) | 0 (0)
Multi organ failure (General disorders) | 1 (1) | 0 (0)
Multi-organ disorder (General disorders) | 0 (0) | 1 (1)
Neck edema (General disorders) | 1 (1) | 0 (0)
Pain aggravated (General disorders) | 1 (1) | 0 (0)
Peripheral edema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Shivering (General disorders) | 8 (9) | 5 (5)
Swelling of legs (General disorders) | 3 (3) | 1 (1)
Swelling of limb (General disorders) | 0 (0) | 1 (1)
Acute liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder edema (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Liver failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 2 (2) | 0 (0)
Bacterial infection due to staphylococcus aureus (Infections and infestations) | 0 (0) | 1 (1)
Bacterial tracheitis (Infections and infestations) | 1 (1) | 3 (3)
Bilateral pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Candida albicans infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Central line infection (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter cloacae infection (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia coli infection (Infections and infestations) | 1 (1) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 4 (4) | 3 (3)
Gram-positive cocci infection (Infections and infestations) | 0 (0) | 1 (1)
Haemophilus influenzae infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes sepsis (Infections and infestations) | 1 (1) | 0 (0)
Infection MRSA (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella pneumoniae infection (Infections and infestations) | 2 (2) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
MRSA (Infections and infestations) | 1 (1) | 0 (0)
Moraxella catarrhalis pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pansinusitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (7) | 3 (3)
Pseudomonas aeruginosa infection NOS (Infections and infestations) | 0 (0) | 1 (1)
Respiratory infection (Infections and infestations) | 15 (19) | 5 (5)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 2 (2)
Rhinovirus infection (Infections and infestations) | 3 (3) | 5 (5)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Septicemia (Infections and infestations) | 0 (0) | 1 (1)
Septicemia due to Escherichia coli (E. coli) (Infections and infestations) | 0 (0) | 1 (1)
Septicemia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Serous otitis media (glue ear) (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcus aureus bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcus aureus cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcus aureus pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Stenotrophomonas maltophilia infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal septicemia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcus pneumoniae pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcus viridans group infection (Infections and infestations) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 2 (2) | 0 (0)
Tracheitis (Infections and infestations) | 3 (3) | 1 (1)
UTI (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 1 (1)
Urine candida (Infections and infestations) | 0 (0) | 1 (1)
Ventilator associated pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Yeast infection (Infections and infestations) | 0 (0) | 1 (1)
Yeast infection of the mouth (Infections and infestations) | 1 (1) | 0 (0)
Abrasions (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Barotrauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bloody airway discharge (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Bruise (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bruise of head (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bruising of hand (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Collapse of lung (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fracture of upper end or unspecified part of radius and ulna, closed (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured cervical spine (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Iatrogenic pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lung injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Renal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin tear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal epidural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALT increased (Investigations) | 1 (1) | 2 (2)
APTT decreased (Investigations) | 0 (0) | 1 (1)
APTT prolonged (Investigations) | 1 (1) | 0 (0)
AST increased (Investigations) | 1 (1) | 4 (5)
Abnormal EEG (Investigations) | 4 (4) | 4 (4)
Albumin decreased (Investigations) | 1 (1) | 0 (0)
Albumin low (Investigations) | 1 (1) | 0 (0)
Amino acid level decreased (Investigations) | 1 (1) | 0 (0)
Amylase high (Investigations) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 4 (4) | 2 (3)
Arterial blood pH decreased (Investigations) | 0 (0) | 1 (1)
Arterial oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
B-type natriuretic peptide (Investigations) | 0 (0) | 1 (1)
BUN increased (Investigations) | 0 (0) | 1 (1)
Bacteria blood identified (Investigations) | 0 (0) | 1 (1)
Band neutrophil count increased (Investigations) | 2 (2) | 1 (1)
Base excess decreased (Investigations) | 1 (1) | 3 (3)
Base excess increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase decreased (Investigations) | 1 (1) | 0 (0)
Blood amino acid level increased (Investigations) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 1 (1)
Blood bicarbonate increased (Investigations) | 1 (1) | 0 (0)
Blood bicarbonate low (Investigations) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood culture positive (Investigations) | 6 (6) | 5 (6)
Blood culture positive viral (Investigations) | 1 (1) | 0 (0)
Blood gases abnormal (Investigations) | 1 (1) | 0 (0)
Blood in urine (Investigations) | 2 (2) | 0 (0)
Blood lactic acid increased (Investigations) | 1 (1) | 0 (0)
Blood osmolarity increased (Investigations) | 0 (0) | 1 (1)
Blood pH abnormal (Investigations) | 0 (0) | 1 (1)
Blood phosphorus increased (Investigations) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Bronchoalveolar lavage abnormal (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
CK increased (Investigations) | 2 (2) | 0 (0)
CO2 total abnormal (Investigations) | 2 (2) | 1 (1)
CPK increase (Investigations) | 0 (0) | 1 (1)
CRP increased (Investigations) | 0 (0) | 1 (1)
Calcium decreased (Investigations) | 1 (1) | 0 (0)
Capillary nail refill test abnormal (Investigations) | 2 (3) | 0 (0)
Carboxyhemoglobin increased (Investigations) | 1 (1) | 0 (0)
Cardiac enzymes increased (Investigations) | 3 (3) | 0 (0)
Cardiac output decreased (Investigations) | 2 (2) | 0 (0)
Chloride increased (Investigations) | 1 (1) | 0 (0)
Chloride low (Investigations) | 0 (0) | 1 (1)
Clotting time increased (Investigations) | 1 (1) | 0 (0)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0)
Cortisol low (Investigations) | 1 (1) | 0 (0)
Creatine kinase increased (Investigations) | 1 (1) | 0 (0)
Creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 2 (3)
Decreased hemoglobin (Investigations) | 2 (2) | 1 (1)
Decreased ventricular afterload (Investigations) | 0 (0) | 1 (1)
Drug level above therapeutic (Investigations) | 0 (0) | 1 (1)
ECG P wave inverted (Investigations) | 1 (1) | 0 (0)
EEG abnormal (Investigations) | 0 (0) | 4 (4)
Elevated liver enzymes (Investigations) | 2 (2) | 1 (1)
End-tidal CO2 decreased (Investigations) | 1 (1) | 0 (0)
Fecal occult blood (Investigations) | 0 (0) | 1 (1)
Function pulmonary decreased (Investigations) | 0 (0) | 1 (1)
Gastric pH decreased (Investigations) | 0 (0) | 1 (1)
Glucose decreased (Investigations) | 1 (1) | 1 (1)
Glucose high (Investigations) | 0 (0) | 2 (2)
Glucose increased (Investigations) | 0 (0) | 1 (1)
Glucose urine present (Investigations) | 0 (0) | 1 (1)
HIE (Investigations) | 1 (1) | 1 (1)
Haemoglobin low (Investigations) | 2 (3) | 4 (4)
Heart rate decreased (Investigations) | 2 (3) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Hematocrit decreased (Investigations) | 1 (1) | 1 (1)
Hematocrit low (Investigations) | 0 (0) | 1 (1)
Hemoglobin decreased (Investigations) | 1 (1) | 1 (1)
INR decreased (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 2 (2)
Increased blood pressure (Investigations) | 1 (1) | 2 (2)
Influenza antibody test positive (Investigations) | 1 (1) | 0 (0)
Ionized calcium decreased (Investigations) | 1 (1) | 1 (1)
LDH decreased (Investigations) | 1 (1) | 0 (0)
LDH increased (Investigations) | 1 (1) | 3 (3)
Lactate dehydrogenase increased (Investigations) | 4 (5) | 6 (6)
Lactate high (Investigations) | 0 (0) | 1 (1)
Lactate increased (Investigations) | 3 (3) | 1 (1)
Lipase increased (Investigations) | 3 (3) | 2 (2)
Liver function tests raised (Investigations) | 1 (1) | 0 (0)
Magnesium decreased (Investigations) | 1 (1) | 1 (1)
Magnesium increased (Investigations) | 1 (1) | 0 (0)
Magnesium low (Investigations) | 1 (1) | 0 (0)
Methicillin-resistant Staphylococcus aureus test positive (Investigations) | 1 (1) | 1 (1)
Neurological examination abnormal (Investigations) | 0 (0) | 1 (1)
Nitrite urine present (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 11 (12) | 8 (8)
PCO2 abnormal (Investigations) | 0 (0) | 1 (1)
PCO2 elevated (Investigations) | 2 (2) | 0 (0)
PCO2 increased (Investigations) | 0 (0) | 1 (1)
PO2 decreased (Investigations) | 1 (1) | 3 (3)
PO2 increased (Investigations) | 1 (1) | 0 (0)
PT increased (Investigations) | 1 (1) | 1 (1)
PTT prolonged (Investigations) | 0 (0) | 1 (1)
Peripheral pulse decreased (Investigations) | 1 (1) | 0 (0)
Phosphate increased (Investigations) | 1 (1) | 0 (0)
Phosphorus low (Investigations) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Potassium decreased (Investigations) | 2 (2) | 5 (5)
Potassium increased (Investigations) | 1 (1) | 1 (1)
Prealbumin (Investigations) | 1 (1) | 0 (0)
Procalcitonin increased (Investigations) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0)
QT prolonged (Investigations) | 3 (3) | 0 (0)
Raised LFTs (Investigations) | 2 (2) | 0 (0)
Respiratory sounds decreased (Investigations) | 1 (1) | 0 (0)
ST segment depression (Investigations) | 1 (1) | 0 (0)
Sodium increased (Investigations) | 1 (1) | 1 (1)
Sodium low (Investigations) | 0 (0) | 2 (2)
Sputum culture positive (Investigations) | 16 (21) | 12 (15)
SvO2 decreased (Investigations) | 1 (1) | 0 (0)
Transaminitis (Investigations) | 3 (3) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 3 (3)
Urine culture positive (Investigations) | 9 (11) | 6 (7)
Urine ketone body present (Investigations) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 7 (8) | 8 (8)
Urine output increased (Investigations) | 1 (1) | 4 (4)
WBC decreased (Investigations) | 3 (3) | 0 (0)
WBC increased (Investigations) | 1 (1) | 1 (1)
pH decreased (Investigations) | 1 (1) | 0 (0)
pH increased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Acidosis metabolic (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Cerebral salt-wasting syndrome (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Feeding difficulties and mismanagement (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperammonemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperamylasemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperchloremia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (16) | 16 (16)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 7 (7)
Hyperlipasemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 12 (12) | 13 (14)
Hyperphosphatemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 15 (15) | 11 (11)
Hypochloremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 11 (11) | 12 (12)
Hypokalemia (Metabolism and nutrition disorders) | 35 (37) | 19 (20)
Hypomagnesemia (Metabolism and nutrition disorders) | 12 (12) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 8 (9) | 8 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (7) | 6 (7)
Hypoproteinemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypovolemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 10 (10) | 3 (4)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Volume overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck rigidity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Twitching of limbs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Weakness in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anoxic brain damage (Nervous system disorders) | 0 (0) | 2 (2)
Autonomic dysfunction (Nervous system disorders) | 0 (0) | 1 (1)
Autonomic instability (Nervous system disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral dysfunction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral edema (Nervous system disorders) | 5 (5) | 3 (3)
Cerebral hematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarct (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischemia (Nervous system disorders) | 0 (0) | 1 (1)
Clonus (Nervous system disorders) | 2 (2) | 1 (1)
Drooling (Nervous system disorders) | 1 (1) | 0 (0)
Dysautonomia (Nervous system disorders) | 1 (1) | 3 (3)
Encephalopathy (Nervous system disorders) | 3 (3) | 1 (1)
Fasciculation (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypertonia (Nervous system disorders) | 2 (2) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic brain damage (Nervous system disorders) | 6 (6) | 2 (2)
Hypoxic encephalopathy (Nervous system disorders) | 3 (4) | 7 (7)
IIIrd nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Increased intracranial pressure (Nervous system disorders) | 0 (0) | 1 (1)
Ischemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Leg spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Memory deficit (Nervous system disorders) | 0 (0) | 1 (1)
Movements abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonic jerks (Nervous system disorders) | 2 (2) | 0 (0)
Myoclonic seizure NOS (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 3 (3) | 1 (1)
Nystagmus (Nervous system disorders) | 2 (2) | 0 (0)
Periventricular leukomalacia (Nervous system disorders) | 1 (1) | 0 (0)
Quadriparesis (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 22 (26) | 14 (15)
Seizures (Nervous system disorders) | 20 (21) | 16 (17)
Shaking (Nervous system disorders) | 2 (2) | 1 (1)
Short-term memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 2 (2) | 3 (3)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Thalamic syndrome (Nervous system disorders) | 9 (9) | 6 (6)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Tremor limb (Nervous system disorders) | 1 (1) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 14 (14) | 5 (5)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Posturing (Psychiatric disorders) | 0 (0) | 3 (3)
Withdrawal syndrome (Psychiatric disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Azotemia (Renal and urinary disorders) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 2 (2) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (2)
Polyuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal function aggravated (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal function disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 4 (4) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Cervix edema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ARDS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acquired tracheobronchomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Airway secretion excessive (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma aggravated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 16 (22)
Bleeding nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Breathing abnormally shallow (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bronchial secretion excessive (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypercarbia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Labored breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal discharge (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pharyngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 11 (13)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 6 (6)
Pulmonary edema recurrent (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Retention carbon dioxide (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Subglottic edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Unspecified disease of respiratory system (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing aggravated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blisters (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Diaper rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Facial swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Macular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Mottled skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pressure sore (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Redness (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin breakdown (Skin and subcutaneous tissue disorders) | 4 (7) | 4 (4)
Skin fissure (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Ulcer skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Acute hypotension (Vascular disorders) | 0 (0) | 2 (2)
Aortic dilatation (Vascular disorders) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 0 (0) | 1 (1)
Clot blood (Vascular disorders) | 0 (0) | 1 (1)
Cold feet (Vascular disorders) | 1 (1) | 0 (0)
Coldness of lower extremities (Vascular disorders) | 0 (0) | 1 (1)
DVT (Vascular disorders) | 1 (1) | 1 (1)
DVT of legs (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis leg (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Flushed (Vascular disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hemodynamic instability (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 16 (17) | 18 (18)
Hypertensive (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 49 (55) | 23 (23)
Hypotension aggravated (Vascular disorders) | 2 (2) | 0 (0)
Hypotensive (Vascular disorders) | 3 (3) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Low blood pressure (Vascular disorders) | 0 (0) | 4 (4)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Poor peripheral perfusion (Vascular disorders) | 1 (1) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 2 (2)
Shock vascular (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis leg (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No